CLINICAL TRIAL: NCT04366726
Title: A Prospective, Single Arm Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Usability of Abaloparatide-sMTS in Postmenopausal Women With Low Bone Mineral Density
Brief Title: Study to Evaluate the Pharmacokinetics (PK), Pharmacodynamics (PD), and Usability of Abaloparatide-solid Microstructured Transdermal System (sMTS) in Postmenopausal Women With Low Bone Mineral Density (BMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BA058-05-022
Record Dates: First submitted 2020-04-16; First posted 2020-04-29 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Postmenopausal Osteoporosis
Keywords: postmenopausal osteoporosis; transdermal delivery; microstructure patch; abaloparatide
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- abaloparatide-sMTS (Experimental): Abaloparatide-sMTS 300 micrograms (μg) was applied to the thigh for 5 minutes once daily for 29 days.
  Interventions: Combination Product: abaloparatide-sMTS

INTERVENTIONS:
Combination Product: abaloparatide-sMTS — Abaloparatide-sMTS is a drug-device combination product consisting of the drug abaloparatide coated onto an sMTS array for transdermal administration of abaloparatide.

SUMMARY:
This was an open-label, single-center study to evaluate the usability of abaloparatide-sMTS by participants with low BMD.

DETAILED DESCRIPTION:
This study aimed to evaluate the ability of participants to self-administer 300 μg abaloparatide-sMTS over a period of 29 days based on PK and PD markers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal for at least 2 years
* BMD T-score based on the female reference range <-1.0 and >-5.0 at the lumbar spine (L1-L4) or hip (femoral neck or total hip) by dual energy X-ray absorptiometry (DXA)
* Good general health as determined by medical history and physical exam (including vital signs, and has a body mass index up to 33 kilograms/square meter (kg/m^2)
* Laboratory tests within the normal range including serum calcium (albumin-corrected), intact parathyroid hormone (PTH), serum phosphorus, alkaline phosphatase, and thyroid stimulating hormone
* Serum 25-hydroxyvitamin D values ≥ 20 nanograms per milliliter (ng/mL)

Exclusion Criteria:

* History of prior external beam or implant radiation therapy involving the skeleton, other than radioiodine
* History of bone disorders other than postmenopausal osteoporosis (such as Paget's disease)
* History of cancer within the last 5 years (with the exception of basal cell or squamous cancer of the skin)
* History of Cushing's disease, hypo or hyperparathyroidism, or malabsorptive syndromes within the past year
* Prior treatment with PTH, PTH-related peptide-derived drugs, or bone anabolic steroids, including abaloparatide, teriparatide, or PTH (1-84)
* Prior treatment with intravenous bisphosphonates at any time or oral bisphosphonates within the past year (12 months). Participants who have received a short course of oral bisphosphonate therapy (3 months or less) may be enrolled as long as the treatment occurred 6 or more months prior to enrollment
* Prior treatment with an investigational drug or device within the past 3 months or 5 half-lives of the investigational drug, whichever is longer

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Radius Health, Inc.
Locations (1):
- Pharmaceutical Research Associates, Inc, Lenexa, Kansas, United States

REFERENCES:
- [Derived] Miller PD, Troy S, Weiss RJ, Annett M, Schense J, Williams SA, Mitlak B. Phase 1b Evaluation of Abaloparatide Solid Microstructured Transdermal System (Abaloparatide-sMTS) in Postmenopausal Women with Low Bone Mineral Density. Clin Drug Investig. 2021 Mar;41(3):277-285. doi: 10.1007/s40261-021-01008-7. Epub 2021 Feb 27. PMID 33638863

RESULTS

PARTICIPANT FLOW:
Groups:
- Abaloparatide-sMTS: Abaloparatide-solid microstructured transdermal system (sMTS) 300 micrograms (μg) was applied to the thigh for 5 minutes once daily for 29 days.
Period: Overall Study
Arm/Group | Abaloparatide-sMTS
Started | 22
Received at Least 1 Dose of Study Drug | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received at least 1 dose of study drug.
Groups:
- Abaloparatide-sMTS: Abaloparatide-sMTS 300 μg was applied to the thigh for 5 minutes once daily for 29 days.
Arm/Group | Abaloparatide-sMTS
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Abaloparatide Maximum Plasma Concentration (Cmax) on Day 29
Time Frame: 0 (predose), 10 minutes, 20 minutes, 30 minutes, 1 hour, 1.5 hours, 2 hours, 3 hours, and 4 hours postdose on Day 29
Population: The Pharmacokinetic Analysis Population included all participants who received at least 1 dose of study drug and who had sufficient evaluable plasma concentrations to reliably estimate 1 or more PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/milliliter (pg/mL)
Arm/Group | Abaloparatide-sMTS
Number analyzed (Participants) | 22
picograms/milliliter (pg/mL) | 399.6 (41.8)

2. Primary Outcome: Abaloparatide Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-t) on Day 29
Time Frame: 0 (predose) and 4 hours postdose on Day 29
Population: The Pharmacokinetic Analysis Population included all participants who received at least 1 dose of study drug and had sufficient evaluable plasma concentrations to reliably estimate 1 or more PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*pg/mL
Arm/Group | Abaloparatide-sMTS
Number analyzed (Participants) | 22
hour*pg/mL | 604.7 (51.1)

3. Secondary Outcome: Percent Change From Baseline of Serum Procollagen Type I N-Terminal Propeptides (s-PINP) at Day 29
Description: Blood samples were taken to measure s-PINP, a bone formation marker. s-PINP concentrations reflect the rate of skeletal new bone formation. Increases in s-PINP indicate anabolic biologic response in the bone.
Time Frame: Baseline, Day 29
Population: The Bone Metabolism Population includes all participants in the Safety Population who have baseline and at least one post-baseline s-PINP.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Abaloparatide-sMTS
Number analyzed (Participants) | 22
percent change | 103.16 (104.729)

4. Secondary Outcome: Change From Baseline of Serum Calcium (Albumin-Corrected) to Predose and Postdose on Day 29
Time Frame: Baseline, 0 (predose) and 4 hours postdose on Day 29
Population: The Safety Population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: millimoles/liter (mmol/L)
Arm/Group | Abaloparatide-sMTS
Number analyzed (Participants) | 22
millimoles/liter (mmol/L)
  Day 29, predose | -0.031 (0.0986)
  Day 29, postdose | -0.002 (0.0659)

5. Secondary Outcome: Change From Baseline of Serum Phosphorus to Predose and Postdose on Day 29
Time Frame: Baseline, 0 (predose) and 4 hours postdose on Day 29
Population: The Safety Population includes all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Abaloparatide-sMTS
Number analyzed (Participants) | 22
mmol/L
  Day 29, predose | 0.051 (0.1832)
  Day 29, postdose | 0.006 (0.1877)

6. Secondary Outcome: Change From Baseline of Cyclic Adenosine Monophosphate (cAMP) to Day 29
Time Frame: Baseline, 0 (predose) and 30-minutes postdose on Day 29
Population: The Safety Population included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: micromoles/liter (μmol/L)
Arm/Group | Abaloparatide-sMTS
Number analyzed (Participants) | 22
micromoles/liter (μmol/L)
  Day 29, predose | -0.0030 (0.0023)
  Day 29, postdose | -0.0006 (0.0046)

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 36
Description: The Safety Population included all participants who received at least 1 dose of study drug.
Groups:
- Abaloparatide-sMTS: Abaloparatide-sMTS was applied to the thigh for 5 minutes once daily for 29 days.
Arm/Group | Abaloparatide-sMTS
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abaloparatide-sMTS (N=22)
Application site erythema (General disorders) | 22
Application site haemorrhage (General disorders) | 6
Application site oedema (General disorders) | 14
Application site pain (General disorders) | 20
Application site pruritus (General disorders) | 6
Application site swelling (General disorders) | 17
Burning sensation (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results may not be published prior to the Study Report completion. Investigators may publish results, providing a manuscript to the Sponsor =/> 30 days prior to its submission to a publisher. Sponsor will provide manuscript to Investigators =/> 30 days prior to its submission. Investigator shall comply with Sponsor's policy, withholding publication for an additional 60 days to permit the Sponsor to obtain patent or other proprietary rights protection, if deemed necessary.

DOCUMENTS (2):
  • Study Protocol (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT04366726/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT04366726/SAP_001.pdf